CLINICAL TRIAL: NCT03372278
Title: Zimmer® Maxera™ Acetabular System in Total Hip Arthroplasty. A Multicenter, Prospective, Non-controlled Post Market Clinical Follow-up Study
Brief Title: PMCF Study on the Safety and Performance of the Zimmer® Maxera™ Acetabular System in Total Hip Arthroplasty
Status: Active, not recruiting | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: CIE2011-01H
Record Dates: First submitted 2017-11-30; First posted 2017-12-13 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Rheumatoid Arthritis With Adequate Bone Quality; Inflammatory Arthritis; Osteoarthritis, Hip; Avascular Necrosis; Post-traumatic; Arthrosis; Congenital Hip Dysplasia
Keywords: Total hip arthroplasty; Medical Device; Safety; Prothesis
MeSH Terms: conditions — Arthritis; Osteoarthritis, Hip; Osteonecrosis; Osteoarthritis; Hip Dislocation, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | US Export: Yes

GROUPS / COHORTS (1):
- Patients who received the Maxera Cup: Subjects in need of a total hip arthroplasty, who met the inclusion/exclusion criteria and who received the Maxera Cup.

SUMMARY:
This study is a multicenter, prospective, non-controlled post market clinical follow-up study. The objectives of this study are to confirm the safety and performance of the commercially available Zimmer® Maxera™ Acetabular System in Total Hip Arthroplasty.

DETAILED DESCRIPTION:
The objectives of this study are to confirm the safety and performance of the Zimmer Maxera Cup mated with either a BIOLOX® delta or BIOLOX® OPTION femoral head when used in primary total hip arthroplasty.

In total 250 patients will be enrolled into the study at up to 10 sites.All potential study subjects will be required to participate in the Informed Consent Process.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 to 75 years of age, inclusive.
* Patient is skeletally mature.
* Patient qualifies for primary unilateral or simultaneous bilateral total hip arthroplasty (THA) based on physical exam and medical history including at least one of the following:

  * Osteoarthritis
  * Avascular necrosis (AVN)
  * Inflammatory arthritis
  * Rheumatoid arthritis with adequate bone quality
  * Post-traumatic arthritis
  * Congenital hip dysplasia.
* Patient has no history of previous total hip replacement or arthrodesis of the affected hip joint(s). Patient has a Harris Hip Score <70 in the affected hip and a Harris Hip pain rating of moderate, marked, or disabled.
* Patient is willing and able to provide written informed consent.
* Patient is willing and able to cooperate in the required post-operative therapy.
* Patient is willing and able to complete scheduled follow-up evaluations as described in the Informed Consent.
* Patient has participated in the Informed Consent process and has signed the Ethics Committee approved informed consent.

Exclusion Criteria:

* The patient is:

  * A prisoner
  * Mentally incompetent or unable to understand what participation in the study entails.
  * A known alcohol or drug abuser
  * Anticipated to be non-compliant
* The patient has a neuromuscular disorder, vascular disorder or other condition that could contribute to prosthesis instability, prosthesis fixation failure, or complications in postoperative care.
* The patient has local bone tumors and/or cysts in the portion of bone to be retained in the operative hip that could inhibit implant fixation.
* The patient has insufficient bone stock or poor bone quality to fix the component. Insufficient bone stock exists in the presence of metabolic bone disease (i.e. osteoporosis), cancer, and radiation. Note: Dual Energy X-ray Absorptiometry (DEXA) may be required to assess the presence of adequate bone stock.
* The patient has rapid disease progression as obvious by joint destruction or bone absorption seen on x-ray.
* The patient has osteoradionecrosis in the affected hip.
* The patient has a neuromuscular condition in the ipsilateral or contralateral limb which affects lower limb function.
* The patient has loss of abductor musculature in the affected hip.
* The patient has a vascular (large and small vessel disease) insufficiency.
* The patient has had previous prosthetic hip replacement device (any type, including surface replacement arthroplasty, endoprosthesis, etc.) in the joint to be operated.
* The patient has had previous girdlestone procedure (resection arthroplasty) or surgical fusion of the hip to be operated.
* The patient has an acute femoral neck fracture in the operative hip.
* The patient has had a procedure on the operative hip in the last 6 months (i.e. arthroscopy, ORIF femoral neck fracture, etc).
* The patient has undergone a total hip replacement, endoprosthesis, or surface arthroplasty of the contralateral (opposite side) hip within the past 6 months regardless of whether the previous hip was enrolled in this clinical study.
* The patient has a moderate to severe limb length discrepancy greater than 3.2 cm.
* The patient has an active, old or remote infection in or about the affected hip joint or an infection distant from the hip joint that may spread to the hip hematogenously.
* The patient has poor skin coverage around the affected hip joint.
* The patient has a diagnosed systemic disease that could affect his/her safety or the study outcome.
* The patient is currently receiving, or within the past three months, has received any drug known to potentially interfere with bone/soft tissue healing (e.g. long-term chronic systemic steroid or inhaler steroid therapy).
* The patient has received an investigational drug or device within the previous 6 months.
* The patient is known to be pregnant.
* The patient is unwilling or unable to give informed consent, or to comply with the followup program.
* The patient is known to have a highly communicable disease that may limit follow-up.
* The patient has a known sensitivity or allergic reaction to one or more of the implanted materials which include metal and ceramic.
* The patient is Grade III obese with a Body Mass Index (BMI) > 35.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from severe hip pain and disability requiring total hip arthroplasty and who meet the inclusion/exclusion criteria
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Implant survival based on removal or intended removal of the device and determined using the Kaplan-Meier method | 10 years post-surgery

SECONDARY OUTCOMES:
Pain and functional performance based on the Harris Hip Score | 10 years post-surgery
Pain and functional performance based on the UCLA Score | 10 years post-surgery
Subject quality-of-life determined by the EQ-5D (EuroQoI) score | 10 years post-surgery
X-rays evaluated for radiolucencies, osteolysis, hypertrophy, subsidence, heterotopic ossification, etc | 10 years post-surgery
Safety based on eventual complications occurred including dislocations and revisions/removals | 10 years post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Achakri, Study Director — Zimmer Biomet
Locations (8):
- The Mater Hospital, Concord Hospital, Sydney, Australia
- UZ Leuven, Pellenberg, Belgium
- Center Maisonneuve-Rosemont Hospital, Montreal, Canada
- Jokilaakson terveys oy, Jämsä, Finland
- Centre Hospitalier de Perpignan, Perpignan, France
- Reinier de Graaf Groep, Delft, Netherlands
- Hospital Son Llatzer, Palma de Mallorca, Spain
- Royal Liverpool and Broadgreen University Teaching Hospitals, Liverpool, United Kingdom